CLINICAL TRIAL: NCT00082524
Title: A Multicenter, Open-Label, Noncomparative Study to Evaluate the Safety, Tolerability, and Efficacy of Caspofungin Acetate in Children With Documented Candida or Aspergillus Infections
Brief Title: Documented Candida or Aspergillus Infections in Pediatric Patients (0991-043)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-043; Formerly-0404CCAI; MK0991-043; 2004_100
Record Dates: First submitted 2004-05-11; First posted 2004-05-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Aspergillosis; Candidiasis
MeSH Terms: conditions — Aspergillosis; Candidiasis | interventions — Caspofungin

INTERVENTIONS:
Drug: caspofungin acetate — Duration of Treatment - 7-90 days
  Other Names: MK0991

SUMMARY:
This study is an open label, noncomparative study using an investigational agent for the treatment of documented Candida or Aspergillus infections in pediatric patients (ages 3 months-17 years).

ELIGIBILITY:
* Children, 3 months through 17 years of age,
* with esophageal candidiasis or
* invasive candidiasis or
* children requiring salvage treatment of invasive aspergillosis.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with one or more drug-related clinical or laboratory adverse experience(s)

SECONDARY OUTCOMES:
The proportion of patients who discontinued due to a drug-related AE or who have a serious drug-related AE
The proportion of patients with a favorable efficacy response to caspofungin therapy in each infection type

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Zaoutis TE, Jafri HS, Huang LM, Locatelli F, Barzilai A, Ebell W, Steinbach WJ, Bradley J, Lieberman JM, Hsiao CC, Seibel N, Laws HJ, Gamba M, Petrecz M, Taylor AF, Strohmaier KM, Chow JW, Kartsonis NA, Ngai AL. A prospective, multicenter study of caspofungin for the treatment of documented Candida or Aspergillus infections in pediatric patients. Pediatrics. 2009 Mar;123(3):877-84. doi: 10.1542/peds.2008-1158. PMID 19255017
- Available data/document: CSRSynopsis — http://www.merck.com/clinical-trials/policies-perspectives.html